The Effect of Logotherapy-Based Intervention on Depression Patients on Depression,
Psychological Pain and Meaning of Life

NCT Number: NCT05702736

Document Date: 2023-08-11

Approved by a Human Subjects Protection Review Board Date: 2020-03-04

**Objectives:** This study aimed to reduce the depressive symptoms and psychological pain levels of the patients and to increase their level of finding meaning in life with the logotherapy intervention applied to patients diagnosed with depression.

**Design and Methods:** A quasi-experimental pre-test, post-test and follow-up test, control group study was conducted. The sample group consisted of depressed patients in a psychiatry department in Izmir. The data were collected for both intervention and control groups in three different time periods: pre-test, post-test and 3-month follow-up. Sixteen of the 48 patients included in the study were excluded because they did not meet the inclusion criteria. The remaining 32 patients were divided into intervention (n = 16) and control group (n = 16). Two patients in the intervention group were excluded for unwilling and two patients were excluded because they could not complete the interviews. As a result, the study was completed with a total of 28 participants, 12 in the intervention group and 16 in the control group. Data collection was conducted simultaneously for the intervention and control groups. Intervention and control groups were contacted by phone for pre-test, post-test (after 8 weeks) and follow-up test (after 3 months) data.